CLINICAL TRIAL: NCT04535193
Title: An Open-Label, Exploratory, Phase 1/2 Scintigraphy Study Evaluating 18F-mFBG for Imaging Myocardial Sympathetic Innervation in Subjects Without and With Heart Disease
Brief Title: Open-Label Study of 18F-mFBG for Imaging Myocardial Sympathetic Innervation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innervate Radiopharmaceuticals LLC (Formerly: Illumina Radiopharmaceuticals LLC) (Industry)
Collaborators: Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP101-121
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases
Keywords: 18F-mFBG; meta-fluorobenzylguanidine
MeSH Terms: conditions — Cardiovascular Diseases | interventions — 3-fluorobenzylguanidine; Administration, Intravenous

STUDY DESIGN:
Intervention Model Description: Study Cohort I will evaluate the myocardial update of 18F-mFBG (as a marker of sympathetic innervation) in control subject with a low likelihood of coronary heart disease.
  Study Cohort II will evaluate the myocardial update of 18F-mFBG (as a marker of sympathetic innervation) in stable patients with heart failure and reduced left ventricular function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low likelihood of coronary heart disease (Other): Thorax and total body imaging for quantification of normal biodistribution and myocardial sympathetic innervation. PET imaging to 210 minutes post-administration.
  Interventions: Drug: 18F-mFBG for intravenous administration
- Heart Failure + left ventricular function (LVEF ≤ 35%) (Other): Thorax and total body imaging for quantification of myocardial sympathetic innervation. PET imaging to 100 minutes post-administration
  Interventions: Drug: 18F-mFBG for intravenous administration

INTERVENTIONS:
Drug: 18F-mFBG for intravenous administration — Positron-emitting tomography (PET) (either PET/CT or PET/MR) imaging agent
  Other Names: meta-fluorobenzylguanidine; IRP101

SUMMARY:
This is a Phase 1/2 study evaluating the positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for quantification of myocardial sympathetic innervation.

DETAILED DESCRIPTION:
This is a Phase 1/2 study evaluating the positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for quantification of myocardial sympathetic innervation. The first part of the study will examine control subjects, patients with very low likelihood of coronary heart disease. This initial part will determine optimal imaging procedures for studying uptake and clearance of 18F-mFBG in myocardial sympathetic neurons and provide preliminary data for estimating radiation dosimetry in adults and developing reference files for quantification of normal and abnormal levels of the radiopharmaceutical. The second part will examine a group of stable patients with New York Heart Association (NYHA) class 2 heart failure (HF) and reduced left ventricular (LV) systolic function (LV ejection fraction (EF) ≤35%). The primary objectives of the second part will be to:

* document the degree to which 18F-mFBG uptake in the heart is reduced and
* characterize the distribution of regional abnormalities in relation to findings on other cardiac imaging studies such as myocardial perfusion (MP) and magnetic resonance (MR) imaging.

Effectiveness of 18F-mFBG will be judged in relation to historical experience with other nuclear imaging agents for cardiac sympathetic innervation imaging such as a 123I-meta-iodobenzylguanidine (mIBG) and 11C-hydroxyephedrine (HED).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at study entry
* able and willing to comply with study procedures
* signed and dated informed consent is obtained
* male or a female who is either surgically sterile (has had a documented bilateral oophorectomy and/or hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom the result of a serum pregnancy test performed at screening is negative.

For control subjects:

* Subject is either:

  * <40 years old and has a likelihood assessment for CAD <10%, or
  * 40-50 years old, has a likelihood assessment for CAD <10%, and a normal stress MPI study or stress echocardiography performed within 6 months before study entry, or
  * Without significant coronary atherosclerotic disease (no arterial stenosis with >30% narrowing) as demonstrated by a coronary angiography performed with 6 months before study entry.

For heart failure subjects:

* Diagnosed with HF at least 1 year before enrollment.
* HF classification NYHA Class II at enrollment.
* Rest left ventricular ejection fraction (LVEF) ≤35% measured by an appropriate method (e.g., radionuclide or contrast ventriculography, ECG-gated SPECT MPI, or echocardiography) within 180 days prior to the study imaging procedure, with no change in clinical condition since the LVEF measurement.
* Primary prevention ICD, implanted at least 6 months before enrollment.
* Clinically stable for at least 30 days before enrollment (e.g., not experiencing continuing chest pain, hemodynamic instability, or clinically significant arrhythmia (including ICD discharge)) and remains stable to the time of the study imaging procedure.

Exclusion Criteria:

* Previously entered into this study or has participated in any other investigational medicinal product or medical device study within 30 days of enrollment.
* History or suspicion of significant allergic reaction or anaphylaxis to any components of the 18F-mFBG imaging agent.
* Ventricular pacemaker that routinely functions (>5% paced beats)
* Cardiac revascularization (e.g., percutaneous transluminal coronary angioplasty, PCI, or CABG), or an acute myocardial infarction within the past 30 days.
* Presents with any other clinically active, serious, life-threatening disease with a life expectancy of less than 1 year or where participation in the study might compromise the management of the subject or other reason that in the judgment of the investigator(s) makes the subject unsuitable for participation in the study.
* Serious non-cardiac medical condition associated with significant elevation of plasma catecholamines including pheochromocytoma.
* Claustrophobic or has a movement disorder that prevents him/her from lying still in a supine position for up to an hour at a time.
* Renal insufficiency (serum creatinine >3.0 mg/dL).
* Use of medications that are known to interfere with uptake of NET-dependent agents and these medications cannot be safely withheld 24 hours before study procedures.
* Participated in a research study using ionizing radiation in the previous 12 months.
* For control subjects: a history of Type I or Type II Diabetes Mellitus, signs/symptoms of neurological disease (e.g., Parkinson's Disease, Multiple System Atrophy, Parkinsonian syndromes), or other diseases known to affect the sympathetic nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Chang in 18F-mFBG uptake | Up to 210 minutes after dosing
  Change in 18F-mFBG uptake in the total body and the normal heart over time (based on serial PET images) to:
  * document the time course of global and regional myocardial activity reflecting specific uptake and clearance of the radiopharmaceutical;
  * estimate individual organ and whole-body radiation dosimetry.
Evaluation of 18F-mFBG for imaging myocardial sympathetic innervation | Up to 100 minutes after dosing
  To demonstrate the extent and degree of global and regional reduced 18F-mFBG myocardial uptake on PET/CT (or PET/MR) of HF subjects with significant LV dysfunction (LVEF≤35%).

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Agarwal, MD, Principal Investigator — Mount Sinai Morningside
Locations (1):
- Mount Sinai Morningside, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No